CLINICAL TRIAL: NCT00962000
Title: Effect of Dialysate Flow Rate on Delivered Dose of Dialysis (Kt/Vurea)
Brief Title: Study of How the Dose of Dialysis is Affected by Dialysate Flow Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: University of Louisville (Other); Vanderbilt University Medical Center (Other); University of California, Davis (Other); Gambro Renal Products, Inc. (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Gambro PI 2009
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease; Chronic Renal Disease
Keywords: Hemodialysis; Dialysis, Renal
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 600 mL/min (Other): Dialysis Flow Rate Start 600mL/min Subject starting dialysis flow rate set at 600mL/min. ABAB sequence where A represents three consecutive dialysis treatments with a dialysate flow rate of 600 mL/min and B represents three consecutive treatments with a dialysate flow rate of 800 mL/min.
  Interventions: Other: Dialysis Flow Rate Start 600mL/min
- 800 mL/min (Other): Dialysis Flow Rate Start 800mL/min Subject starting dialysis flow rate set at 800mL/min. BABA sequence where B represents three consecutive treatments with a dialysate flow rate of 800 mL/min and A represents three consecutive dialysis treatments with a dialysate flow rate of 600 mL/min.
  Interventions: Other: Dialysis Flow Rate Start 800mL/min

INTERVENTIONS:
Other: Dialysis Flow Rate Start 600mL/min — ABAB sequence where A represents three consecutive dialysis treatments with a dialysate flow rate of 600 mL/min and B represents three consecutive treatments with a dialysate flow rate of 800 mL/min.
  Arms: 600 mL/min
Other: Dialysis Flow Rate Start 800mL/min — BABA sequence where B represents three consecutive treatments with a dialysate flow rate of 800 mL/min and A represents three consecutive dialysis treatments with a dialysate flow rate of 600 mL/min.
  Arms: 800 mL/min

SUMMARY:
The purpose of this study is to look at how the dose of dialysis is affected by the rate at which dialysate flows through the dialyzer. The dose of dialysis (Kt/V) will be determined by measuring blood levels of urea at the beginning and end of dialysis at two different dialysate flow rates.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject ≥18 years of age undergoing chronic hemodialysis for end- stage renal disease (ESRD) three times a week for at least three months with a stable treatment prescription
* Subject has no hospitalizations in previous three months for a significant illness related to a renal or dialysis problem except for vascular access surgery
* Subject with an AV fistula or graft capable of routinely delivering a blood flow rate of 400 mL/min

Exclusion Criteria:

* Subject who is non-compliant with dialysis prescription
* Subject whose hemodialysis schedule is not three times a week
* Subject using a catheter for blood access
* Subject who is not anticoagulated with heparin during hemodialysis
* Subject with a current malignancy involving sites other than skin
* Subject with a history of drug or alcohol abuse within the last six months
* Subject who is believed to be unable to complete the entire study (e.g., due to a concurrent disease, life expectancy of less than a year, or scheduled kidney transplant
* Subject who is pregnant
* Subject who is considered incompetent to give an informed consent
* Subject with a positive test for hepatitis B surface antigen within the past 30 days (testing for hepatitis B surface antigen is not required for subjects who have tested positive for hepatitis B antibody within the past year and any such patients will not be subject to this exclusion criterion)
* Subject with known HIV infection (if this is not known, no HIV testing will be performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ward, Ph.D., Principal Investigator — University of Louisville
Locations (3):
- United States (3):
  - University of California Davis, Sacramento, California
  - University of Louisville, Louisville, Kentucky
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Background] Daugirdas JT. Second generation logarithmic estimates of single-pool variable volume Kt/V: an analysis of error. J Am Soc Nephrol. 1993 Nov;4(5):1205-13. doi: 10.1681/ASN.V451205. PMID 8305648
- [Background] Daugirdas JT, Schneditz D. Overestimation of hemodialysis dose depends on dialysis efficiency by regional blood flow but not by conventional two pool urea kinetic analysis. ASAIO J. 1995 Jul-Sep;41(3):M719-24. doi: 10.1097/00002480-199507000-00107. PMID 8573901

RESULTS

PARTICIPANT FLOW:
Groups:
- 600 mL/Min First: Subject starting dialysis flow rate set at 600mL/min. Following an ABAB study design where A represents three consecutive dialysis treatments with a dialysate flow rate of 600 mL/min and B represents three consecutive treatments with a dialysate flow rate of 800 mL/min.
- 800 mL/Min First: Subject starting dialysis flow rate set at 800mL/min. Following an BABA study design where B represents three consecutive dialysis treatments with a dialysate flow rate of 800 mL/min and A represents three consecutive treatments with a dialysate flow rate of 600 mL/min.
Period: Period 1 - 1 Week
Arm/Group | 600 mL/Min First | 800 mL/Min First
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Period 2 - 1 Week
Arm/Group | 600 mL/Min First | 800 mL/Min First
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Period 3 - 1 Week
Arm/Group | 600 mL/Min First | 800 mL/Min First
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Period 4 - 1 Week
Arm/Group | 600 mL/Min First | 800 mL/Min First
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All subjects who participated in the study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 42
Age, Continuous [Mean (Full Range); unit: years]
  >=18 years | 50 [19 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 26
Pre-dialysis Weight [Mean (Full Range); unit: kg] | 84 [48 to 147]

OUTCOME MEASURES:

1. Primary Outcome: Delivered Single-pool Kt/Vurea (spKt/V) at Dialysate Flow Rates of 600 mL/Min and 800 mL/Min.
Description: The dose of dialysis delivered in a single treatment is commonly expressed in terms of Kt/Vurea, where K is the clearance of urea, t is the treatment time, and V is the urea distribution volume. When urea is removed from a single compartment during dialysis, it is called the "single-pool" Kt/V. Delivered Kt/Vurea was determined from pre-and post-dialysis BUN concentrations measured during the final treatment session of each group (ABAB or BABA).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: single-pool Kt/Vurea (spKt/V)
Units Other Than Participants: Treatments
Groups:
- 600 mL/Min: Dialysate flow rate of 600 mL/min
- 800 mL/Min: Dialysate flow rate of 800 mL/min
Arm/Group | 600 mL/Min | 800 mL/Min
Number analyzed (Participants) | 42 | 42
Number analyzed (Treatments) | 75 | 77
single-pool Kt/Vurea (spKt/V) | 1.66 (0.25) | 1.63 (0.21)
Statistical Analysis 1: Comparison: 600 mL/Min vs 800 mL/Min; Increasing the dialysate flow rates from 600 mL/min to 800 mL/min will not significantly increase Kt/Vurea; Test type: Non-Inferiority or Equivalence — The sample size required for the study was estimated using a web-based power calculation tool. Analysis of data from some 50,000 hemodialysis patients showed a within-patient between-treatment standard deviation of 0.21 for Kt/Vurea. Using this estimate of standard deviation, 38 subjects would be needed to detect a difference in Kt/Vurea of 0.1 with a significance level of 0.05 and a power of 90% with two determinations per subject at each level of dialysate flow rate; ANOVA — There is no p values because the power calculation is based on the primary outcome variable; The three centers and the two flow rates were treated as fixed effects and the subjects within centers modeled as a random effect; Mean Difference (Final Values) = -0.024, 95% CI 2-sided [-0.064 to 0.024], Standard Error of Mean 0.02217

2. Secondary Outcome: Delivered Equilibrated Kt/Vurea (eKt/V at Dialysate Flow Rates of 600 mL/Min and 800 mL/Min.
Description: The dose of dialysis delivered in a single treatment is commonly expressed in terms of Kt/Vurea, where K is the clearance of urea, t is the treatment time, and V is the urea distribution volume. The formula for equilibrated Kt/Vurea takes urea rebound into consideration. Delivered Kt/Vurea was determined from pre-and post-dialysis BUN concentrations measured during the final treatment session of each group (ABAB or BABA).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: equilibrated Kt/Vurea (eKt/V)
Units Other Than Participants: Treatments
Arm/Group | 600 mL/Min | 800 mL/Min
Number analyzed (Participants) | 42 | 42
Number analyzed (Treatments) | 75 | 77
equilibrated Kt/Vurea (eKt/V) | 1.37 (0.20) | 1.35 (0.18)
Statistical Analysis 1: Comparison: 600 mL/Min vs 800 mL/Min; Increasing the dialysate flow rates from 600 mL/min to 800 mL/min will not significantly increase Kt/Vurea; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — There is no p value for eKt/V because the power calculation is based on the primary outcome variable (Kt/Vsp) alone; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.014, 95% CI 2-sided [-0.051 to 0.023], Standard Error of Mean 0.01849

3. Secondary Outcome: Kt/V Determined From Measurements of Ionic Dialysance
Description: Kt/VID was determined for all study treatments at 2 of the 3 centers using on-line clearance measurements (Gambro Diascan or Fresenius On-line Clearance Monitor).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Kt/VID
Units Other Than Participants: Treatments
Arm/Group | 600 mL/Min | 800 mL/Min
Number analyzed (Participants) | 28 | 28
Number analyzed (Treatments) | 140 | 143
Kt/VID | 1.46 (0.24) | 1.49 (0.35)
Statistical Analysis 1: Comparison: 600 mL/Min vs 800 mL/Min; Increasing the dialysate flow rates from 600 mL/min to 800 mL/min will not significantly increase Kt/Vurea; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — There is no p value for Kt/VID because the power calculation is based on the primary outcome variable (Kt/Vsp) alone; Mean Difference (Final Values) = 0.035, 95% CI [-0.029 to 0.099], Standard Error of Mean 0.03103

ADVERSE EVENTS:
Arm/Group | 600 mL/Min First | 800 mL/Min First
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days